CLINICAL TRIAL: NCT03881475
Title: Validation of an Early Detection Questionnaire of Burnout in Healthcare Workers at Clermont-Ferrand University Hospital
Brief Title: Early Detection of Burnout - Healthcare Workers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: CHU-432
Record Dates: First submitted 2019-03-08; First posted 2019-03-19 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Healthcare Workers; Stress; Occupation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthcare workers: Participants will participate in several sessions where they will complete the questionnaires. The questionnaires will be spaced: 0, 1 week, 6 months, 1 year and then at each occupational visit within 5 years.
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — During consultations in occupational medicine (periodic visit and / or visit at the request of the employee), the nurses (or physicians) will propose the passation of the questionnaire to the voluntary agents.
  The questionnaire, composed of 79 items with 2 validated questionnaires (HAD and MBI), will be filled using a digital tablet (via the REDCAP software).
  Time required to complete the questionnaire 10 minutes.

SUMMARY:
Burnout is a public health issue. Healthcare workers are particularly at risk of burnout with occupational stress identified as the major risk factor. The "Health Work Environment" service is composed of physicians, nurses and psychologist with the aim of providing efficient and adapted care for healthcare workers at CHU of Clermont-Ferrand. In addition, they must ensure a role of primary, secondary and tertiary prevention. With regard to burnout, the majority of the work carried out concerns tertiary prevention, that is to say the care of a person in a situation of burnout. It would be necessary to carry out secondary prevention in order that people at risk of burnout can be detected earlier. However, there is currently no individual questionnaire to detect early burnout

DETAILED DESCRIPTION:
Early detection of burnout was designed to provide a better understanding of warning sign of burnout in order to detect earlier workers at risk.

In the present protocol, parameters are measured on several occasions (0, 1 week, at 6 month, at 12 months and then at each occupational visit within 5 years).

Statistical analysis will be performed using Stata software (version 13; Stata-Corp, College Station, Tex., USA). All statistical tests will be two-sided and p<0.05 will be considered significant. After testing for normal distribution (Shapiro-Wilk test), data will be treated either by parametric or non-parametric analyses according to statistical assumptions. Inter-groups comparisons will systematically be performed 1) without adjustment and 2) adjusting on factors liable to be biased between groups.

Analysis will be performed using anova or Kruskal-Wallis (KW) tests. When appropriate (p<0.05), a post-hoc test for multiple comparisons (Tukey-Kramer after anova and Dunn post KW) will be used.

Comparisions of categorical variables will be performed using Chi-squared or Fischer test. Marascuillo's procedure will be performed for multiple comparisons. Relations between quantitative outcomes will be analyzed using correlation coefficients (Pearson or Spearman). Fisher's Z transformation and William's T2 statistic will be performed to compare correlations between variables and within a single group of subjects. Longitudinal data will be treated using mixt-model analyses in order to treat fixed effects group, time and group x time interaction taking into account between and within participant variability.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers at Clermont-Ferrand Hospital
* Aged: from 18 years to retirement

Exclusion Criteria:

* Participant refusal to participate
* No healthcare workers at Clermont-Ferrand Hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workers at Clermont-Ferrand Hospital
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Level of burnout, anxiety and depression. | at day 1
  To assess the ability of a questionnaire of early detection of burnout, two validated questionnaires will be used: Maslach Burnout Inventory - Human Service Survey (in order to measure level of burnout) and Hospital Anxiety Depression Scale (in order to measure the presence of anxious or depressive symptoms).
  No other psychological or physiological measures will be taken.
Level of anxiety | at day 1
  To assess the ability of a questionnaire of early detection of burnout, two validated questionnaires will be used: Maslach Burnout Inventory - Human Service Survey (in order to measure level of burnout) and Hospital Anxiety Depression Scale (in order to measure the presence of anxious or depressive symptoms).
  No other psychological or physiological measures will be taken.
Level of depression | at day 1
  To assess the ability of a questionnaire of early detection of burnout, two validated questionnaires will be used: Maslach Burnout Inventory - Human Service Survey (in order to measure level of burnout) and Hospital Anxiety Depression Scale (in order to measure the presence of anxious or depressive symptoms).
  No other psychological or physiological measures will be taken.

CONTACTS AND LOCATIONS:
Overall Officials: Frederic DUTHEIL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France